CLINICAL TRIAL: NCT05086276
Title: A Phase 2, Prospective, Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Multicenter Study to Evaluate the Efficacy of FX-322 Administered by Intratympanic Injection in Adults With Acquired Sensorineural Hearing Loss
Brief Title: FX-322 in Adults With Acquired Sensorineural Hearing Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Frequency Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX-322-208
Record Dates: First submitted 2021-10-08; First posted 2021-10-20 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Hearing Loss, Sensorineural; Noise Induced Hearing Loss; Sudden Hearing Loss
Keywords: Intratympanic administration; Restoration of hearing loss
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Noise-Induced; Hearing Loss, Sudden

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FX-322 (Active Comparator): FX-322, 1 dose
  Interventions: Drug: FX-322
- Placebo (Placebo Comparator): Placebo, 1 dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FX-322 — Active Comparator
  Arms: FX-322
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2, prospective, randomized, double-blind, placebo-controlled, single-dose, multicenter study to evaluate the efficacy of FX-322, administered by intratympanic injection, in adults with acquired sensorineural hearing loss (SNHL).

DETAILED DESCRIPTION:
This is a Phase 2, prospective, randomized, double-blind, placebo-controlled, single-dose, multicenter study to evaluate the efficacy of FX-322, administered by intratympanic injection, in adults with acquired sensorineural hearing loss (SNHL).

Previous human studies in subjects 18 to 65 years inclusive (FX-322-103, FX-322-201, FX-322-111) and subjects 66-85 inclusive (FX-322-112) demonstrated that a single dose FX-322 was well tolerated in patients with acquired SNHL with no treatment-related serious adverse events. Adverse events in these studies were generally common to and associated with the intratympanic injection procedure with mild and transient discomfort in patients both with the drug and the placebo.

Frequency Therapeutics' Investigators intend to evaluate efficacy with a single dose of FX-322 in subjects 18 to 65 years inclusive with acquired SNHL.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has read and voluntarily signed the Informed Consent Form (ICF) after all questions have been answered and prior to any study-mandated procedure.
2. Adult aged 18-65 years inclusive at Screening.
3. Documented medical history consistent with acquired, adult onset, sensorineural hearing loss associated with noise-induced SNHL (NIHL) or idiopathic sudden SNHL (SSNHL) (documented audiogram at least 6 months prior to screening required).
4. A pure tone average at the Screening Visit of 35-85 dB at 500Hz, 1000Hz, 2000Hz, and 4000Hz in the ear to be injected.
5. Ability to communicate well with the Investigator and is willing to comply with and complete all the study procedures.
6. Female subjects must be of non-childbearing potential or will need to utilize two methods of highly effective contraception during the study participation (e.g. hormonal contraception and condom or an intrauterine device and condom) or remain abstinent. Male subjects should use condoms with spermicide during the course of the study or remain abstinent. Subjects should not donate sperm or ova during the study period.
7. Have met additional masked criteria as determined by the Electronic Data Capture system.

Exclusion Criteria:

1. Subject has previously been randomized in a FX-322 clinical trial.
2. Perforation of tympanic membrane or other tympanic membrane disorders that would interfere with the delivery and safety assessment of an intratympanic medication or reasonably be suspected to affect tympanic membrane healing after injection in study ear. This includes a current tympanostomy tube.
3. Any conductive hearing loss of greater than 15 dB at a single frequency or greater than 10dB at two or more contiguous octave frequencies in the study ear at the Screening visit.
4. Active chronic middle ear disease or a history of major middle ear surgery, as an adult, in the ear to be injected.
5. Subject has had an intratympanic injection in either ear within 3 months of the screening visit.
6. Evidence of or previous diagnosis of auditory neuropathy, traumatic brain injury, "central" hearing loss, or genetic hearing loss.
7. History of chronic, recurrent clinically significant vestibular symptoms.
8. History of bilateral sudden sensorineural hearing loss or recurrent sudden sensorineural hearing loss.
9. History of clinically significant systemic autoimmune disease (e.g. rheumatoid arthritis, Sjogren's syndrome, multiple sclerosis, psoriasis).
10. History of head or neck radiation, treatment, or exposure to platinum based chemotherapy drugs or aminoglycosides.
11. Exposure to another investigational drug within 28 days prior to screening visit.
12. Evidence of any active or chronic disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would pose an unacceptable risk to the subject in the opinion of the investigator following a detailed medical history, physical examination, and vital signs (systolic and diastolic blood pressure, pulse rate, body temperature).
13. Positive urine pregnancy test or breast-feeding.
14. Any known factor, condition, or disease that, in the view of the Investigator, might interfere with treatment compliance, study conduct or interpretation of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Director — Frequency Therapeutics
Locations (26):
- United States (26):
  - Clinical Trial Site, Tucson, Arizona
  - Clinical Trial Site, Fresno, California
  - Clinical Trial Site, Torrance, California
  - Clinical Trial Site, Colorado Springs, Colorado
  - Clinical Trial Site, Sarasota, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Marrero, Louisiana
  - Clinical Trial Site, Novi, Michigan
  - Clinical Trial Site, Omaha, Nebraska
  - Clinical Trial Site, Albany, New York
  - Clinical Trial Site, Amherst, New York
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Oklahoma City, Oklahoma
  - Clinical Trial Site, Charleston, South Carolina
  - Clinical Trial Site, Orangeburg, South Carolina
  - Clinical Trial Site, Spartanburg, South Carolina
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Fort Worth, Texas
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Murray, Utah
  - Clinical Trial Site, St. George, Utah
  - Clinical Trial Site, Norfolk, Virginia
  - Clinical Trial Site, Richmond, Virginia
  - Clinical Trial Site, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- FX-322: Single intratympanic injection of FX-322 (laduviglusib 0.628 mg/sodium valproate 17.72 mg) into affected ear
- Placebo: Single intratympanic injection of placebo into affected ear
Period: Overall Study
Arm/Group | FX-322 | Placebo
Started | 70 | 72
Completed | 69 | 71
Not Completed | 1 | 1
Not completed — Missed visit 5/Day 60 visit | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set is defined as the subjects who met all inclusion criteria who received at least 1 dose of study drug. Note that 2 subjects who received FX-322 treatment were ultimately not included in the Full Analysis Set because, after they had been treated and as study assessments progressed, they were deemed to not meet the inclusion criteria for sensorineural hearing loss (SNHL) and were excluded from the FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | FX-322 | Placebo | Total
Number analyzed (Participants) | 68 | 72 | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.9 (11.12) | 50.6 (12.20) | 51.7 (11.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 29 | 45
  Male | 52 | 43 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 61 | 63 | 124
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 60 | 64 | 124
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 68 | 72 | 140

OUTCOME MEASURES:

1. Primary Outcome: Word Recognition in Quiet
Description: Percent of subjects exceeding the Carney-Schlauch 95% confidence interval for improvement from baseline in number of words recognized from Consonant-Nucleus-Consonant (CNC) word lists
Time Frame: Baseline through Day 90
Population: Full Analysis Set is defined as all randomized subjects that met inclusion criteria who received one dose of study drug
Measure: Number; unit: Percent of subjects
Arm/Group | FX-322 | Placebo
Number analyzed (Participants) | 68 | 72
Percent of subjects | 14.7 | 11.1
Statistical Analysis 1: Comparison: FX-322 vs Placebo; Test type: Superiority; p = 0.525, Chi-squared — P value for statistical significance is <0.05; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.51 to 3.73]
Statistical Analysis 2: Comparison: FX-322 vs Placebo; Test type: Superiority; p = 0.525, Chi-squared — P value for statistical significance is <0.05; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [-7.52 to 14.71]

2. Secondary Outcome: Words-in-Noise
Description: Mean absolute percent change in number of recognized words from CNC word lists
Time Frame: Baseline through Day 90
Population: Full Analysis Set is defined as all randomized subjects that met inclusion criteria who received one dose of study drug
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | FX-322 | Placebo
Number analyzed (Participants) | 67 | 72
Percent change | 0.17 (2.465) | 0.35 (3.295)
Statistical Analysis 1: Comparison: FX-322 vs Placebo; Test type: Superiority; p = 0.973, Mixed Models Analysis — P value for statistical significance is <0.05; Least squares mean difference = 0.02, 95% CI 2-sided [-0.954 to 0.987], Standard Error of Mean 0.491

3. Secondary Outcome: Standard Pure Tone Audiometry
Description: Mean overall pure tone average (PTA) hearing thresholds in decibels (dB) derived by averaging the air conduction thresholds at 0.5, 1, 2 and 4 kHZ frequencies
Time Frame: Baseline through Day 90
Population: Full Analysis Set is defined as all randomized subjects that met inclusion criteria who received one dose of study drug
Measure: Mean (Standard Deviation); unit: Decibels (dB)
Arm/Group | FX-322 | Placebo
Number analyzed (Participants) | 68 | 72
Decibels (dB) | 65.09 (7.865) | 63.91 (9.816)

4. Secondary Outcome: Patient Global Impression of Change (PGI-C) Hearing Loss Scale
Description: Average response in PGI-C hearing loss scale, using the assigned numeric values of 1-5: 1) much better, 2) a little better, 3) no change, 4) a little worse 5) much worse
Time Frame: Day 90
Population: Full Analysis Set is defined as all randomized subjects that met inclusion criteria who received one dose of study drug
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | FX-322 | Placebo
Number analyzed (Participants) | 68 | 71
Score on a scale | 3.0 (0.52) | 2.9 (0.64)
Statistical Analysis 1: Comparison: FX-322 vs Placebo; Test type: Superiority; p = 0.160, ANCOVA — P value for statistical significance is <0.05; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.06 to 0.34], Standard Error of Mean 0.10

5. Secondary Outcome: Patient Global Impression of Change (PGI-C) Daily Impacts Scale
Description: Average response in PGI-C daily impacts scale, using the assigned numeric values of 1-5: 1) much better, 2) a little better, 3) no change, 4) a little worse 5) much worse
Time Frame: Day 90
Population: Full Analysis Set is defined as all randomized subjects that met inclusion criteria who received one dose of study drug
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | FX-322 | Placebo
Number analyzed (Participants) | 68 | 71
Score on a scale | 3.0 (0.53) | 2.8 (0.60)
Statistical Analysis 1: Comparison: FX-322 vs Placebo; Test type: Superiority; p = 0.027, ANCOVA — P value for statistical significance is <0.05; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [0.03 to 0.41], Standard Error of Mean 0.10

ADVERSE EVENTS:
Time Frame: Baseline through Day 90
Description: Safety analysis set (SAS) is defined as subjects that received at least one dose of study drug.The SAS includes the two subjects not included in the FAS that did not meet inclusion criteria for SNHL but were dosed with drug.
Arm/Group | FX-322 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/72
Serious Adverse Events (participants affected / at risk) | 1/70 | 1/72
Other Adverse Events (participants affected / at risk) | 41/70 | 44/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FX-322 (N=70) | Placebo (N=72)
Device-related infection (Infections and infestations) | 0 | 1 — One subject experienced a device-related infection, pneumonia parainfluenzae viral, sepsis, and encephalopathy. These SAEs were not deemed related to the study drug
Encephalopathy (Nervous system disorders) | 0 | 1
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Extragonadal primary seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — One subject developed a seminoma during the trial period. This was not deemed related to the study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FX-322 (N=70) | Placebo (N=72)
Audiogram abnormal (Investigations) | 16 | 22
Blood pressure increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1
Drug screen positive (Investigations) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 8 | 7
Ear pain (Ear and labyrinth disorders) | 3 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 4
Ear discomfort (Ear and labyrinth disorders) | 2 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 2 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0
Myringosclerosis (Ear and labyrinth disorders) | 1 | 0
Ototoxicity (Ear and labyrinth disorders) | 1 | 0
Injection site pain (General disorders) | 13 | 7
Injection site scab (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Injection site discomfort (General disorders) | 1 | 0
Injection site hemorrhage (General disorders) | 1 | 0
Edema (General disorders) | 0 | 1
COVID-19 (Infections and infestations) | 5 | 7
Bronchitis (Infections and infestations) | 2 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Candida infection (Infections and infestations) | 1 | 0
Device-related infection (Infections and infestations) | 0 | 1
Ear injection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Pneumonia parainfluenze viral (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2
Seizure (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Hyperammonemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Blepharospasm (Eye disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0
Extragonadal primary seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Decreased interest (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Feeling of despair (Psychiatric disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs must obtain sponsor's written consent before publishing or presenting the trial results

DOCUMENTS (2):
  • Study Protocol (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT05086276/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT05086276/SAP_001.pdf